CLINICAL TRIAL: NCT01792856
Title: Randomized Controlled Trial on Recovery-oriented Coaching Intervention for Patients With Early Psychosis
Brief Title: Coaching Intervention for Patients With Early Psychosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Eric Y H Chen, Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UW 12-486
Record Dates: First submitted 2013-01-31; First posted 2013-02-15 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Schizophrenia
Keywords: coaching; early psychosis; schizophrenia
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- intervention group (Experimental): Subjects are scheduled to receive a 6-month group-based recovery-oriented coaching program. This is a structured, manualised treatment program based on life coaching principles with cognitive-behavioural and solution-focused elements incorporated. It guides subjects to undergo an active, yet stepwise change process by stimulating motivation, setting achievable goals, generation of action plans via collaborative exploration, fostering self-regulatory capacity, and provision of autonomy-supportive treatment environment and peer support. Subjects' perceived competence, sense of control, self-management skills and hence functioning will be improved via successful experiences and positive feelings generated after attainment of self-initiated goals. Cognitive-behavioural techniques such as self-monitoring, activity scheduling and behavioural modification will be employed.
  Interventions: Other: Recovery-oriented intervention
- control group (Experimental): Subjects will receive group-based supportive therapy provided by case managers of JCEP project. The therapy provides patients with psychoeducation about psychosis, stress management, emotional and social support. Coaching and cognitive-behavioural techniques will not be incorporated. Therapy sessions and duration will be comparable to that of recovery-oriented coaching program.
  Interventions: Other: psychoeducation

INTERVENTIONS:
Other: Recovery-oriented intervention — Life coaching is defined as a collaborative, solution-focused, outcome-oriented and systematic process which aims to facilitate enhancement of life experience and goal attainment of an individual in various life domains. It is based on the theoretical framework of positive psychology and behavioural change model, and targets at building up an individual's potential via fostering hope, motivation, self-efficacy and self-regulation. The principles of life coaching thus closely align with recovery orientation that emphasizes on self-initiation and empowerment via person-centred and strength-based approach.
  Other Names: Life-coaching approach
  Arms: intervention group
Other: psychoeducation — Subjects will receive group-based supportive therapy provided by case managers of JCEP project. The therapy provides patients with psychoeducation about psychosis, stress management, emotional and social support. Coaching and cognitive-behavioural techniques will not be incorporated. Therapy sessions and duration will be comparable to that of recovery-oriented coaching program.
  Other Names: Control group
  Arms: control group

SUMMARY:
Jockey Club Early Psychosis (JCEP) project is a territory-wide specialized EI service that is launched in August 2009 and provides 3-year phase-specific intervention for adult patients presenting with first-episode psychosis (FEP) to psychiatric units of Hospital Authority (HA). To promote early functional recovery, JCEP project develops recovery-oriented intervention based on life coaching approach (recovery-oriented coaching) in addition to case management. This is a structured group-based coaching program incorporating cognitive-behavioural and solution-focused therapeutic components. The program facilitates patients to undergo active change process via identification of achievable goals, formulation of action plans, provision of feedback and progress monitoring for goal attainment. Subjects will be randomized (block size: 2) to receive either recovery-oriented coaching program (intervention group) or supportive therapy (control group).

Intervention group Subjects are scheduled to receive a 6-month group-based recovery-oriented coaching program. This is a structured, manualised treatment program based on life coaching principles with cognitive-behavioural and solution-focused elements incorporated. It guides subjects to undergo an active, yet stepwise change process by stimulating motivation, setting achievable goals, generation of action plans via collaborative exploration, fostering self-regulatory capacity, and provision of autonomy-supportive treatment environment and peer support. Subjects' perceived competence, sense of control, self-management skills and hence functioning will be improved via successful experiences and positive feelings generated after attainment of self-initiated goals. Cognitive-behavioural techniques such as self-monitoring, activity scheduling and behavioural modification will be employed.

Control group Subjects will receive group-based supportive therapy provided by case managers of JCEP project. The therapy provides patients with psychoeducation about psychosis, stress management, emotional and social support. Coaching and cognitive-behavioural techniques will not be incorporated. Therapy sessions and duration will be comparable to that of recovery-oriented coaching program.

Assessments Each subject will be assessed at three time points, i.e., baseline before randomization (T1), 12 weeks (T2, post-phase I intervention) and 24 weeks (T3, post-phase II intervention). Assessments on symptomatology, functioning and subjective wellbeing will be administered at all time points. Cognitive and reinforcement learning assessments will be conducted at T1 and T3. functional magnetic resonance imaging (fMRI) will be performed at T1 and T3 for the first 20 subjects recruited in each treatment group. A group of healthy volunteers matched in sex, age and educational level will be recruited from the community with fMRI, cognitive and reinforcement learning evaluations done at T1 and T3. To maintain blinding to treatment assignment, assessments will be conducted by research assistants who are independent of treatment delivery and randomization. Subjects will be trained to not reveal their treatment allocation before each follow-up assessment.

DETAILED DESCRIPTION:
Background, current evidence and key references

Psychotic disorders including schizophrenia are severe mental illnesses that affect 3% of the population and constitute an enormous burden to patients and the society. They cause profound disruptions in patients' functioning including independent living skills, relationships, scholastic and vocational development, and are ranked by World Health Organization as the third most disabling medical condition. In an attempt to minimize long-term disability, numerous early intervention (EI) programs for psychosis have been established worldwide in the past decade. It is based on the premise that shortening of treatment delay and provision of phase-specific treatments in the initial few years of psychosis can improve illness outcome. Literature indicated that patients who received EI had better clinical and functional outcomes than those treated by standard psychiatric care. Nonetheless, accumulating evidence has suggested that a significant proportion of early psychosis patients exhibited functional deterioration even in the presence of clinical remission. Studies have also consistently shown that patients with psychosis frequently experience motivational deficits and diminished goal-directed behaviours which are key negative symptoms predictive of functional outcome. Functional disability thus represents an unmet therapeutic need in EI for psychosis.

In this regard, there is a shift of therapeutic focus from symptom control to functional enhancement. It is also increasingly recognized that patients' perspectives should be taken into consideration in conceptualizing functional recovery and developing recovery-oriented service to further improve functional outcome . Owing to lack of effective treatments in addressing functional impairment, recently, there is an emerging interest in adopting life coaching to complement other interventions by its specific focus on motivation and functioning. Life coaching is defined as a collaborative, solution-focused, outcome-oriented and systematic process which aims to facilitate enhancement of life experience and goal attainment of an individual in various life domains . It is based on the theoretical framework of positive psychology and behavioural change model, and targets at building up an individual's potential via fostering hope, motivation, self-efficacy and self-regulation. The principles of life coaching thus closely align with recovery orientation that emphasizes on self-initiation and empowerment via person-centred and strength-based approach. In fact, empirical evidence suggested that hopelessness and low self-efficacy were associated with poor functioning in early psychosis. Conversely, increased motivation was shown to enhance both functional and cognitive outcomes in schizophrenia . Additionally, studies evaluating coaching in non-clinical population found that it significantly improved subjects' motivation and psychological wellbeing. Despite the growing recognition and adoption of life coaching approach in mental health services, it has rarely been applied in the early course of psychotic disorder.

Jockey Club Early Psychosis (JCEP) project is a territory-wide specialized EI service that is launched in August 2009 and provides 3-year phase-specific intervention for adult patients presenting with first-episode psychosis (FEP) to psychiatric units of Hospital Authority (HA). To promote early functional recovery, JCEP project develops recovery-oriented intervention based on life coaching approach (recovery-oriented coaching) in addition to case management. This is a structured, group-based coaching program incorporating cognitive-behavioural and solution-focused therapeutic components. The program facilitates patients to undergo active change process via identification of achievable goals, formulation of action plans, provision of feedback and progress monitoring for goal attainment. Unlike the majority of therapies that focus mainly on symptoms and functional deficiencies, this program is strength-oriented and aims to facilitate patients to gain a sense of agency and to achieve sustained functional improvement via firstly, enhancing motivation, self-regulation and competence by positive reinforcement obtained from successive accomplishments of self-determined goals; secondly, providing an autonomy-supportive treatment environment with a context of recovery expectations; and thirdly, facilitating formation of supportive social network in group-based setting.

We have previously examined perceptions of early psychosis patients on recovery, with achievement of adequate functioning being regarded as a key element signifying recovery. Our earlier study on FEP patients with EI revealed that less than one-fifth achieved recovery and only 43% of remitted patients were in functional remission at the end of 3-year follow-up. Thus, in line with the literature, our findings indicated an urgent need for developing effective interventions to optimize patients' functional outcome in the early illness stage which is otherwise regarded as a critical window of opportunity for minimizing long-term disability. In this context, recovery-oriented coaching program which specifically addresses motivational and functional impairments may prove to be an effective psychosocial intervention for promoting functional recovery, and thereby worthy of systematic evaluation in patients with early psychosis.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnostic and Statistical Manual (DSM)-IV diagnosis of schizophrenia, schizoaffective disorder, schizophreniform disorder, delusional disorder or brief psychotic disorder;
2. 26 to 64 years;
3. illness duration <5 years;
4. positive symptoms of mild or lower severity (rating <4 in all items of Positive Symptom Subscale of PANSS);
5. impaired functioning with SOFAS score <=60;
6. Cantonese speaking.

Exclusion Criteria:

* substance abuse
* organic psychotic disorders and
* mental retardation

Ages: 25 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2013-02; Primary Completion 2015-02 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Social functioning | 24 weeks
  Social Functioning will be measured by Social and Occupational Functioning Assessment Scale (SOFAS) and Role Functioning Scale and Occupational Life Functioning Scale and Social Functioning Scale (SFS).
  Vocational status will be obtained.
  To evaluate the efficacy of recovery-oriented coaching, a series of analysis of variance (ANOVAs) are used to test the significance of differences between intervention and control groups at 12 weeks and 24 weeks on social functioning.
Negative Symptoms (esp.intrinsic motivation) | 24weeks
  Positive and Negative Syndrome Scale (PANSS) and Scale for the Assessment of Negative Symptoms (SANS) will be used to assess negative symptoms.
  Intrinsic motivation is evaluated using the sum of 3 items from Quality of Life Scale i.e., sense of purpose, motivation and curiosity.
  A series of analysis of variance (ANOVAs) are used to test the significance of differences between intervention and control groups at 12 weeks and 24 weeks on negative symptoms and Intrinsic motivation

SECONDARY OUTCOMES:
Subjective Wellbeing | 24 weeks
  Quality of Life (SF-12), state hope scale , chinese general self-efficacy scale and Rosenberg self-esteem scale will be used to evaluate subjective wellbeing of patients.
  A series of analysis of variance (ANOCAs) are used to test the significance of differences between intervention and control groups at 12 weeks and 24 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Wing Chung Chang, Dr., Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, China

REFERENCES:
- [Background] van Os J, Kapur S. Schizophrenia. Lancet. 2009 Aug 22;374(9690):635-45. doi: 10.1016/S0140-6736(09)60995-8. PMID 19700006
- [Background] World Health Organization. World Health Report 2001: mental health: new understanding, new hope. Geneva: WHO; 2001.
- [Background] McGlashan TH. Early detection and intervention of schizophrenia: rationale and research. Br J Psychiatry Suppl. 1998;172(33):3-6. PMID 9764119
- [Background] Harvey PO, Lepage M, Malla A. Benefits of enriched intervention compared with standard care for patients with recent-onset psychosis: a metaanalytic approach. Can J Psychiatry. 2007 Jul;52(7):464-72. doi: 10.1177/070674370705200709. PMID 17688011
- [Background] Robinson DG, Woerner MG, McMeniman M, Mendelowitz A, Bilder RM. Symptomatic and functional recovery from a first episode of schizophrenia or schizoaffective disorder. Am J Psychiatry. 2004 Mar;161(3):473-9. doi: 10.1176/appi.ajp.161.3.473. PMID 14992973
- [Background] Chang WC, Tang JY, Hui CL, Lam MM, Chan SK, Wong GH, Chiu CP, Chen EY. Prediction of remission and recovery in young people presenting with first-episode psychosis in Hong Kong: a 3-year follow-up study. Aust N Z J Psychiatry. 2012 Feb;46(2):100-8. doi: 10.1177/0004867411428015. PMID 22311526
- [Background] Foussias G, Remington G. Negative symptoms in schizophrenia: avolition and Occam's razor. Schizophr Bull. 2010 Mar;36(2):359-69. doi: 10.1093/schbul/sbn094. Epub 2008 Jul 21. PMID 18644851
- [Background] Bellack AS. Scientific and consumer models of recovery in schizophrenia: concordance, contrasts, and implications. Schizophr Bull. 2006 Jul;32(3):432-42. doi: 10.1093/schbul/sbj044. Epub 2006 Feb 3. PMID 16461575
- [Background] Bora R, Leaning S, Moores A, Roberts G. Life coaching for mental health recovery: the emerging practice of recovery coaching. Adv Psychiatr Treat 2010; 16:459-467.
- [Background] Grant AM. The impact of life coaching on goal attainment, megacognition and mental health. Soc Behav Personal 2003; 31:253-264.
- [Background] Pratt SI, Mueser KT, Smith TE, Lu W. Self-efficacy and psychosocial functioning in schizophrenia: a mediational analysis. Schizophr Res. 2005 Oct 15;78(2-3):187-97. doi: 10.1016/j.schres.2005.02.014. PMID 16154054
- [Background] Nakagami E, Hoe M, Brekke JS. The prospective relationships among intrinsic motivation, neurocognition, and psychosocial functioning in schizophrenia. Schizophr Bull. 2010 Sep;36(5):935-48. doi: 10.1093/schbul/sbq043. Epub 2010 May 12. PMID 20462998
- [Background] Green LS, Oades LG, Grant M. Cognitive-behavioral, solution-focused life coaching: enhancing goal striving, wellbeing, and hope. J Positive Psychology 2006; 1:142-149.
- [Background] Lam MM, Pearson V, Ng RM, Chiu CP, Law CW, Chen EY. What does recovery from psychosis mean? Perceptions of young first-episode patients. Int J Soc Psychiatry. 2011 Nov;57(6):580-7. doi: 10.1177/0020764010374418. Epub 2010 Jul 5. PMID 20603266